CLINICAL TRIAL: NCT04258969
Title: Evaluating the Feasibility of Pedaling at a Low-moderate Intensity During Chemotherapy Infusions in Colorectal Cancer Patients.
Brief Title: Pedaling at a Low-Moderate Intensity During Chemotherapy Administration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19101113
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Exercise, Aerobic; Chemotherapy; Chemotherapeutic Toxicity
Keywords: Pedaling; Sarcopenia; Quality of Life
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pedaling Group (Experimental): During the first 2 hours of their chemotherapy infusions, participants will pedaling for 30 minutes using a stationary cycle ergometer. Participants will be allowed to determine their pedaling intensity and cadence, however, will be encouraged to reach the established goal intensity level. Additionally, subjects will complete both a physical activity questionnaire (International Physical Activity Questionnaire) and a quality of life questionnaire (European Organization for Research and Treatment of Cancer QLQ - CR 29) at baseline and following their last chemotherapy treatment. A questionnaire on chemotherapy side effects (Memorial Symptom Assessment Scale) will be gathered at baseline, during chemotherapy cycles 3, 6, and/or 12, and following completion of chemotherapy treatment. Lastly, muscular strength and physical performance will be measured via grip strength tests and TGUG tests within 2-4 weeks of the post-surgery and chemotherapy completion CT scans.
  Interventions: Behavioral: Pedaling

INTERVENTIONS:
Behavioral: Pedaling — Participants will pedaling at a low-moderate intensity using a stationary pedal ergometer concurrent to their chemotherapy (FOLFOX or FOLFIRI) infusion. Participants will cycle for 30 min within the first 2 hours of their infusion.

SUMMARY:
The purpose of this study is to evaluate the feasibility of completing a low-moderate intensity pedaling session concurrent to chemotherapy treatment for colorectal cancer. Secondary objectives for this study consist of evaluating the role of pedaling on sarcopenia rates, quality of life markers, chemotherapy side effects, rate of hospital admissions, and treatment delays.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed colon or rectal cancer with previous surgical intervention and planned intravenous chemotherapy treatment (FOLFOX or FOLFIRI).
* ECOG Performance Status of Grade 0-2.

Exclusion Criteria:

* Limited functional status, demonstrated by an ECOG Performance Status of Grade 3-5.
* Severe cardiac history or comorbidities (i.e. have a cardiac defibrillator or have a history of heart failure, clinically significant aortic stenosis, cardiac arrest, uncontrolled angina, uncontrolled arrhythmias, major heart surgery, stroke, or pulmonary embolus).
* Chest pain or severe shortness of breath at rest or with physical activity.
* Orthopedic impediments to exercise (i.e. joint immobility or lower extremity lymphedema).
* Limitations to sustained exercise (i.e. bone metastases in the femur neck).
* Severe arthritis (i.e. osteoarthritis or rheumatoid arthritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of Pedaling Concurrent to Chemotherapy Infusion | 12-24 weeks
  The number of completed pedaling sessions as well as the ability of patients to meet goal pedaling intensities will be evaluated.

SECONDARY OUTCOMES:
Quality of Life Scores | 12-24 weeks
  Quality of life markers will be assessed using the European Organization for Research and Treatment of Cancer [EORTC] QLQ - CR 29 at baseline and following their last chemotherapy treatment.
Sarcopenia Rates | 12-24 weeks
  The presence of sarcopenia is best defined by evaluating muscle mass, muscle strength, and physical performance. CT scans will be obtained at time of diagnosis (pre-surgery), post-surgery (pre-chemotherapy), and following chemotherapy completion. Patient's CT scans will be uploaded to a medical image analysis software (SliceOmatic) which allows for the evaluation of body composition. Within 2-4 weeks of the post-surgery and chemotherapy completion CT scans, muscular strength and physical performance will be measured via grip strength tests and Timed- Get-Up and Go tests, respectively.
Hospital Admission Rates | 12-24 weeks
  The number of hospital admissions during chemotherapy timeframe will be evaluated.
Symptom Severity | 12-24 weeks
  A questionnaire on chemotherapy side effects (Memorial Symptom Assessment Scale) will be gathered at baseline, during chemotherapy cycles 3, 6, and/or 12, and following completion of chemotherapy treatment to measure severity of chemotherapy-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Hayden, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States